CLINICAL TRIAL: NCT06475625
Title: Clinical Impact of Orsiro™ Stent in Patient With Chronic Kidney Disease Undergoing Percutaneous Coronay Intervention : A Multicenter, Prospective All-comers Registry
Brief Title: Clinical Impact of Orsiro™ Stent in Patient With Chronic Kidney Disease
Acronym: OKAY
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Mahn-Won Park, Professor, The Catholic University of Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC190OEDI0069
Record Dates: First submitted 2024-06-18; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases; Coronary Artery Disease
Keywords: Chronic Kidney Diseases; Coronary Artery Disease; Orsiro stent
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal or mild renal dysfunction (Experimental): eGFR ≥ 60 ml·min - 1·1.73㎡
  Interventions: Procedure: Percutaneous coronary intervention; Device: Orsiro™ or Orsiro_Mission™ stent
- Moderate renal dysfunction (Experimental): 30≤ eGFR< 60 ml·min - 1·1.73㎡
  Interventions: Procedure: Percutaneous coronary intervention; Device: Orsiro™ or Orsiro_Mission™ stent
- Severe renal dysfunction (Experimental): eGFR < 30 ml·min -1·1.73㎡
  Interventions: Procedure: Percutaneous coronary intervention; Device: Orsiro™ or Orsiro_Mission™ stent

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention
Device: Orsiro™ or Orsiro_Mission™ stent — Percutaneous coronary intervention with Orsiro™ or Orsiro_Mission™ stents

SUMMARY:
Orsiro™ or Orsiro_Mission™ stents have the biodegradable polymer and the thinnest stent strut (60㎛) in commercially available stents, which could minimize chronic inflammation and incomplete endothelialization. In several prior studies, ultrathin strut sirolimus-eluting stent (Orsiro®) showed better outcomes in terms of target lesion failure or target lesion revascularization compared to other contemporary stents. Chronic kidney disease (CKD) is known to be associated with adverse cardiovascular outcome including restenosis or stent thrombosis following percutaneous coronary interventin (PCI), because the patients with CKD have more complex coronary lesion characteristics, severe calcification, and diffuse plaque of the coronary artery. However, there is a paucity of data regarding clinical efficacy of Orsiro® in CKD population. Therefore, this study aims to investigate the differences in clinical outcomes according to renal function in patients undergoing PCI with Orsiro™ or Orsiro_Mission™ stents. After patients will be divided into three groups according to the renal function; normal or mild renal dysfunction (eGFR ≥ 60 ml·min - 1·1.73㎡), moderate renal dysfunction ( 30≤ eGFR< 60 ml·min - 1·1.73㎡), and severe renal dysfunction (eGFR < 30 ml·min -1·1.73㎡), the clinical outcome will be investigated among groups.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Patient undergoing percutaneous coronary intervention with Orsiro™ or Orsiro_Mission™ stents

Exclusion Criteria:

* Patient with a life expectancy of less than one year
* Patient who used another drug-eluting stent for percutaneous coronary intervention at study registration time
* Cardiogenic shock
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3113 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Target-lesion failure (TLF) | Within one year after the intervention
  Number of participants with Target-lesion failure (TLF), defined as composite of cardiac death, target vessel-related myocardial infarction (TVMI) and ischemia-driven target-lesion revascularization (TLR) at 1 year

SECONDARY OUTCOMES:
Number of participants with all cause death | Within three years after the intervention
Number of participants with cardiac death | Within three years after the intervention
Number of participants with myocardial infarction | Within three years after the intervention
  periprocedural or spontaneous
Number of participants with composite of death or myocardial infarction | Within three years after the intervention
Number of participants with composite of cardiac death or myocardial infarction | Within three years after the intervention
Number of participants with target-vessel revascularization | Within three years after the intervention
Number of participants with target-lesion revascularization | Within three years after the intervention
Number of participants with stent thrombosis | Within three years after the intervention
  Stent thrombosis appropriate for Academic Research Consortium criteria
Number of participants with target-vessel failure | Within three years after the intervention
  composite of composite of death, nonfatal myocardial infarction and ischemia-drive target-vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Mahn-Won Park, Study Chair — Daejeon St. Mary's Hospital , The Catholic University of Korea
Locations (1):
- Daejeon St. Mary's Hospital , The Catholic University of Korea, Daejeon, South Korea